CLINICAL TRIAL: NCT03274375
Title: Prospective Assessment of Efficacy of Immunoadsorption Therapy in Managing Childhood NMDA-Receptor (NMDAR) Antibodies Encephalitis
Brief Title: Immunoadsorption Therapy in Managing NMDAR Antibodies Encephalitis
Acronym: IANMDAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150919; 2016-A00259-42 (Other: IDRCB)
Record Dates: First submitted 2017-07-24; First posted 2017-09-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Anti-NMDAR Encephalitis
Keywords: Anti-NMDAR encephalitis; IA adsorption; Paediatric
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IA session (Experimental): * 4 Rituximab injections
  * 10 IA sessions
  Interventions: Drug: IA session; Drug: Rituximab

INTERVENTIONS:
Drug: IA session — 10 IA sessions performed in 28 days maximum, using TherasorbTM adsorbers which contain sheep derived polyvalent antihuman-immunoglobulin coupled to SepharoseTM CL-4B.
Drug: Rituximab — Concomitantly, Rituximab will be given each week for 4 weeks (one injection by week +/- 3 days):
  * at least 1 day before each IA session
  * the last injection will occur after the last session IA (minimum one day after)

SUMMARY:
The purpose of the study is to assess the efficacy of immunoadsorption therapy (IA) on improving the neurological status of severe pediatric anti-NMDAR encephalitis patients.

DETAILED DESCRIPTION:
Anti-NMDA-Receptor (NMDAR) encephalitis, the most frequent autoimmune encephalitis after Acute Demyelinating encephalomyelitis (ADEM), affects children with predominant movement disorders, decline of consciousness, psychiatric symptoms, language dysfunction, seizures, dysautonomic symptoms. The cerebrospinal fluid (CSF) is most often abnormal with lymphocytic pleocytosis, CSF-specific oligoclonal bands with intrathecal synthesis of anti-NMDAR antibodies. Antibody titres in CSF and serum seem correlated with clinical outcome. Early start of immunotherapy has been reported to improve clinical outcome and associated with less relapses. In a recent large series (211 children/577), 77% of the patients were admitted to Intensive Care Unit (ICU) at the beginning. Within the group of children, first-line immunotherapy (95%) consisted of corticosteroids (89%), and/or intravenous immunoglobulins (IgIV) (83%), and/or plasma exchange (28%) with failure in 46%. The second-line immunotherapy consisting in rituximab (24%) and/or cyclophosphamide (16%) was proposed in 32%, and tended to be associated with good outcome (OR=3.35, CI: 0.86-12.98, p=0.081 for 53 children; statistical significance was achieved for the entire population including adults (OR: 2.69, CI: 1.24-5.80, p = 0.012) and less relapses.

In investigators' experience, the clinical benefit of rituximab is delayed over one month, while children go on worsening (50% admitted in ICU) thus claiming for faster removal of the antibodies. Plasma exchange is proposed in most of the series as alternative or combined treatment in the acute stage (first-line immunotherapy); recently, another plasmatherapy, immunoadsorption therapy (IA), has been reported as an efficient therapeutic approach in 11/13 patients. In this retrospective study, patients received a median of 6 IA sessions within a median period of 8 days with relevant clinical improvement. However these encouraging results and investigators' experience in few children need further prospective and standardized evaluation.

In IANMDAR study, each patient will receive 10 IA sessions during 28 days maximum. Rituximab will be given each week for 4 weeks (one injection by week +/- 3 days):

* at least 1 day before each IA session
* the 4 injections should be done before V2 (Day 28 after the inclusion)

To assess the efficacy of IA-therapy at short term, the neurological status of patients will be evaluated before and after the 10 IA sessions using the Pediatric Cerebral Performance Category Scale (PCPCS) and the modified Rankin Scale (mRS).

To assess the efficacy of IA-therapy at long term, patients will have a standardized follow-up during two years including neuropsychological evaluation at 1 year and at 2 years (see below for further details).

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-18 years inclusive
* Autoimmune encephalitis with positive anti-NMDAR antibodies in CSF (definite anti-NMDAR encephalitis according to Graus's criteria (Graus et al., 2016).
* PCPCS and mRS at 4 or over at the inclusion after first line therapy (steroids and/or IgIV) when Rituximab therapy is warranted
* Parents or legal guardians signed the Informed consent form
* Social insurance affiliation

Exclusion Criteria:

* Autoimmune encephalitis without NMDAR antibodies
* PCPCS and mRS scores under 4 after first-line therapy
* Contraindication to perform central vascular access
* Pregnancy, breastfeeding or absence of effective contraception (including abstinence) in a pubertal patient.
* Contraindication to perform IA therapy :

  * Clinical conditions that prohibit transitory volume changes
  * Indications that prohibit anticoagulation using Heparin and/or ACD-A solutions
  * History of hypercoagulability
  * Generalized viral, bacterial and/or mycotic infections
  * Severe immune deficiencies (e.g. AIDS)
  * Suspected allergies against sheep antibodies or agarose

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Neurological status evaluated with the Pediatric Cerebral Performance Category Scale (PCPCS) | before and after the 10 IA sessions, 28 days maximum
  at least reduction of 1 point in PCPCS between the two evaluations is expected
Change in Neurological status evaluated with the modified Rankin Scale (mRS) | before and after the 10 IA sessions, 28 days maximum
  at least reduction of 1 point in mRS between the two evaluations is expected

SECONDARY OUTCOMES:
Need of hospitalization in ICU and pediatric neurology unit | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Duration of hospitalization in ICU and pediatric neurology unit | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Need for mechanical ventilation | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Need for vasopressive treatment | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Time of recovery of independent daily-life activities | 28 days
  independent ambulation, enteral feeding, responsiveness to simple instructions and verbal communication (first word)
Name and duration of medication for behavioral disorders and sleep disorders | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Evolution of movement disorders assessed by the Movement Disorder Childhood Scale with video-taping, performed before and after IA therapy | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Biological evolution of NMDAR antibodies tested in serum | 28 days
  before and after IA sessions
Biological evolution of NMDAR antibodies tested in CSF | 28 days
  at diagnosis and after IA sessions
Titration of NMDAR antibodies in serum before and after the first and the last (tenth) IA session | 28 days
  To assess immunoadsorption therapy at short term in pediatric severe anti-NMDAR encephalitis patients
Duration of each immunoadsorption treatment | 28 days
  To assess tolerance of IA therapy
Duration of use of medication for sedation by pharmaceutical class | 28 days
  to assess need of sedation
Occurrence of hypotension with need for vasopressive treatment | 28 days
  To assess tolerance of IA therapy
Occurrence of dysautonomic events (linked to the pathology): cardiac arrhythmia and heart rate events, flush, apnea | 28 days
  To assess tolerance of IA therapy
Occurrence of vascular access complications : Infections (number, duration of antibiotics used), inadvertent removal, inefficiency (duration of retention of each vascular access) | 28 days
  To assess tolerance of IA therapy
Total duration of the immunoadsorption therapy | 28 days
  To assess tolerance of IA therapy
Total number of sessions | 28 days
  To assess tolerance of IA therapy
Number of adsorbers used for each patient | 28 days
  To assess tolerance of IA therapy
Adverse events of associated treatments | 28 days
  To assess tolerance of IA therapy
PCPCS score | 3 months
  To assess Immunoadsorption therapy at long term
mRS score | 3 months
  To assess Immunoadsorption therapy at long term
PCPCS score | 6 months
  To assess Immunoadsorption therapy at long term
mRS score | 6 months
  To assess Immunoadsorption therapy at long term
PCPCS score | 1 year
  To assess Immunoadsorption therapy at long term
PCPCS score | at 2 years
  To assess Immunoadsorption therapy at long term
mRS score | 1 year
  To assess Immunoadsorption therapy at long term
mRS score | at 2 years
  To assess Immunoadsorption therapy at long term
Need of hospitalization in functional rehabilitation unit | 2 years
  To assess Immunoadsorption therapy at long term
Duration of hospitalization in functional rehabilitation unit | 2 years
  To assess Immunoadsorption therapy at long term
School attendance (special school or not) and rehabilitation attendance | 2 years
  To assess Immunoadsorption therapy at long term
Neuropsychological assessment for cognitive and behavioral status with Wechsler scales | 1 year
Neuropsychological assessment for cognitive and behavioral status with Wechsler scales | at 2 years
Neuropsychological assessment for cognitive and behavioral status with Child Behavior Checklist (CBCL) | 1 year
Neuropsychological assessment for cognitive and behavioral status with Child Behavior Checklist (CBCL) | at 2 years
Neuropsychological assessment for cognitive and behavioral status with Brief Inventory of Executive Functions (BRIEF) | 1 year
Neuropsychological assessment for cognitive and behavioral status with Brief Inventory of Executive Functions (BRIEF) | at 2 years
Neuropsychological assessment for cognitive and behavioral status with Pediatric Quality of Life questionnaire (PedsQL) | 1 year
Neuropsychological assessment for cognitive and behavioral status with Pediatric Quality of Life questionnaire (PedsQL) | at 2 years
Visual attention evaluated with NEPSY scale | 1 year
Visual attention evaluated with NEPSY scale | at 2 years
Rey's figure test to evaluate visuospatial abilities and memory | 1 year
Rey's figure test to evaluate visuospatial abilities and memory | 2 years
CMS to assess memory | 1 year
CMS to assess memory | 2 years
Digit span to assess memory | 1 year
Digit span to assess memory | 2 years
Movement disorders assessment with the Movement Disorder Childhood Scale | 3 months
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with video-taping | 3 months
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with the Movement Disorder Childhood Scale | 6 months
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with video taping | 6 months
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with the Movement Disorder Childhood Scale | 1 year
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with the Movement Disorder Childhood Scale | 2 years
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with video-taping | 1 year
  To assess Immunoadsorption therapy at long term
Movement disorders assessment with video-taping | at 2 years
  To assess Immunoadsorption therapy at long term
Occurrence and date of relapses | 2 years
Presence of NMDAR antibodies in CSF | 6 months
  titration at 6 months
Presence of NMDAR antibodies in CSF | 1 year
  titration at 1 year
Presence of NMDAR antibodies in serum | 3 months
  titration at 3 months
Presence of NMDAR antibodies in serum | 6 months
  titration at 6 months
Presence of NMDAR antibodies in serum | 1 year
  titration at 1 year
Proteinorachia | 6 months
  titration at 6 months
Proteinorachia | 1 year
  titration at 1 year
Presence of oligoclonal bands in serum | 1 year
  checked at 1 year
Presence of oligoclonal bands in serum | 3 months
  checked at 3 months
Presence of oligoclonal bands in serum | 6 months
  checked at 6 months
Presence of oligoclonal bands in CSF | 6 months
  checked at 6 months
Presence of oligoclonal bands in CSF | 1 year
  checked at 1 year
Number of lymphocytes in serum | 3 months
  checked at 3 months
Number of lymphocytes in serum | 6 months
  checked at 6 months
Number of lymphocytes in serum | 1 year
  checked at 1 year
Number of lymphocytes in CSF | 6 months
  checked at 6 months
Number of lymphocytes in CSF | 1 year
  checked at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rémi SALOMON, Md, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants-Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No